CLINICAL TRIAL: NCT02911090
Title: Endometriosis Pelvic Pain Interdisciplinary Cohort (EPPIC) Data Registry
Brief Title: Endometriosis Pelvic Pain Interdisciplinary Cohort Data Registry
Acronym: EPPIC
Status: Enrolling by invitation | Type: Observational
Sponsor: BC Women's Hospital & Health Centre (Other)
Collaborators: UBC Department of Obstetrics and Gynaecology (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Paul Yong, Research Director, BC Women's Hospital & Health Centre
Other Study IDs: H16-00264
Record Dates: First submitted 2016-08-31; First posted 2016-09-22 (Estimated); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Endometriosis
Keywords: Endometriosis; Chronic pelvic pain; Dyspareunia
MeSH Terms: conditions — Endometriosis; Dyspareunia | interventions — Routinely Collected Health Data

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Data Registry — Data Registry

SUMMARY:
The purpose of this data registry is to prospectively collect data from patients referred to an interdisciplinary clinic for pelvic pain and endometriosis to investigate long-term patient outcomes, prognosis, predictors, causes, and treatment of pelvic pain and endometriosis.

DETAILED DESCRIPTION:
The BC Women's Centre for Pelvic Pain and Endometriosis is the tertiary referral centre for endometriosis/pelvic pain in British Columbia, Canada. The Centre offers a unique interdisciplinary approach including minimally invasive surgery, hormonal and other medical therapy, pain education, physiotherapy, and CBT/mindfulness.

After informed consent, patients prospectively consent to data collection in the online registry. The registry consists of patient intake questionnaires (including validated measures), physical and ultrasound examination, review of medical records, surgical findings, and annual outcomes to 5 years.

The online data registry is housed in the Research Electronic Data Capture (REDCap) platform located at BC Children's Hospital.

ELIGIBILITY:
Inclusion Criteria:

* All new and re-referred patients at the BC Women's Centre for Pelvic Pain and Endometriosis.

Exclusion Criteria:

* Patients at the BC Women's Centre for Pelvic Pain and Endometriosis seen for reasons other than chronic pelvic pain and/ or endometriosis as well as patients who decline to complete the online questionnaire.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients at the BC Women's Centre for Pelvic Pain and Endometriosis seen for chronic pelvic pain and/ or endometriosis
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Patient-reported severity of chronic pelvic pain | 3 months
  Measured on a scale of 0 (no pain) to 10 (worst pain imaginable)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Yong, MD PhD FRCSC, Principal Investigator — BC Women's Hospital & Health Centre
Locations (1):
- BC Women's Hospital & Health Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Orr NL, Wahl KJ, Lisonek M, Joannou A, Noga H, Albert A, Bedaiwy MA, Williams C, Allaire C, Yong PJ. Central sensitization inventory in endometriosis. Pain. 2022 Feb 1;163(2):e234-e245. doi: 10.1097/j.pain.0000000000002351. PMID 34030173
- [Background] McPeak AE, Allaire C, Williams C, Albert A, Lisonkova S, Yong PJ. Pain Catastrophizing and Pain Health-Related Quality-of-Life in Endometriosis. Clin J Pain. 2018 Apr;34(4):349-356. doi: 10.1097/AJP.0000000000000539. PMID 28731958
- [Background] Bao C, Noga H, Allaire C, Williams C, Bedaiwy MA, Sadownik LA, Brotto LA, Smith KB, Yong PJ. Provoked Vestibulodynia in Women with Pelvic Pain. Sex Med. 2019 Jun;7(2):227-234. doi: 10.1016/j.esxm.2019.03.002. Epub 2019 Apr 4. PMID 30954496
- [Background] Ng N, Wahl K, Orr NL, Noga H, Williams C, Allaire C, Bedaiwy MA, Yong PJ. Endometriosis and Negative Perception of the Medical Profession. J Obstet Gynaecol Can. 2020 Mar;42(3):248-255. doi: 10.1016/j.jogc.2019.08.034. Epub 2019 Dec 18. PMID 31864912
- [Background] Williams C, Long AJ, Noga H, Allaire C, Bedaiwy MA, Lisonkova S, Yong PJ. East and South East Asian Ethnicity and Moderate-to-Severe Endometriosis. J Minim Invasive Gynecol. 2019 Mar-Apr;26(3):507-515. doi: 10.1016/j.jmig.2018.06.009. Epub 2018 Jun 20. PMID 29935381
- [Background] Arion K, Orr NL, Noga H, Allaire C, Williams C, Bedaiwy MA, Yong PJ. A Quantitative Analysis of Sleep Quality in Women with Endometriosis. J Womens Health (Larchmt). 2020 Sep;29(9):1209-1215. doi: 10.1089/jwh.2019.8008. Epub 2020 Mar 13. PMID 32176592
- [Background] Geoffrion R, Yang EC, Koenig NA, Brotto LA, Barr AM, Lee T, Allaire C, Bedaiwy MA, Yong PJ. Recreational Cannabis Use Before and After Legalization in Women With Pelvic Pain. Obstet Gynecol. 2021 Jan 1;137(1):91-99. doi: 10.1097/AOG.0000000000004207. PMID 33278297
- [Background] Orr NL, Huang AJ, Liu YD, Noga H, Bedaiwy MA, Williams C, Allaire C, Yong PJ. Association of Central Sensitization Inventory Scores With Pain Outcomes After Endometriosis Surgery. JAMA Netw Open. 2023 Feb 1;6(2):e230780. doi: 10.1001/jamanetworkopen.2023.0780. PMID 36848090
- [Background] Shum LK, Bedaiwy MA, Allaire C, Williams C, Noga H, Albert A, Lisonkova S, Yong PJ. Deep Dyspareunia and Sexual Quality of Life in Women With Endometriosis. Sex Med. 2018 Sep;6(3):224-233. doi: 10.1016/j.esxm.2018.04.006. Epub 2018 May 22. PMID 29801714
- [Background] Orr NL, Noga H, Williams C, Allaire C, Bedaiwy MA, Lisonkova S, Smith KB, Yong PJ. Deep Dyspareunia in Endometriosis: Role of the Bladder and Pelvic Floor. J Sex Med. 2018 Aug;15(8):1158-1166. doi: 10.1016/j.jsxm.2018.06.007. PMID 30078464
- [Background] Tucker DR, Noga HL, Lee C, Chiu DS, Bedaiwy MA, Williams C, Allaire C, Talhouk A, Yong PJ. Pelvic pain comorbidities associated with quality of life after endometriosis surgery. Am J Obstet Gynecol. 2023 Aug;229(2):147.e1-147.e20. doi: 10.1016/j.ajog.2023.04.040. Epub 2023 May 4. PMID 37148956
- [Result] Yosef A, Allaire C, Williams C, Ahmed AG, Al-Hussaini T, Abdellah MS, Wong F, Lisonkova S, Yong PJ. Multifactorial contributors to the severity of chronic pelvic pain in women. Am J Obstet Gynecol. 2016 Dec;215(6):760.e1-760.e14. doi: 10.1016/j.ajog.2016.07.023. Epub 2016 Jul 18. PMID 27443813
- [Result] Yong PJ, Williams C, Bodmer-Roy S, Ezeigwe C, Zhu S, Arion K, Ambacher K, Yosef A, Wong F, Noga H, Britnell S, Yager H, Bedaiwy MA, Brotto LA, Albert AY, Lisonkova S, Allaire C. Prospective Cohort of Deep Dyspareunia in an Interdisciplinary Setting. J Sex Med. 2018 Dec;15(12):1765-1775. doi: 10.1016/j.jsxm.2018.10.005. Epub 2018 Nov 13. PMID 30446474
- [Result] Allaire C, Williams C, Bodmer-Roy S, Zhu S, Arion K, Ambacher K, Wu J, Yosef A, Wong F, Noga H, Britnell S, Yager H, Bedaiwy MA, Albert AY, Lisonkova S, Yong PJ. Chronic pelvic pain in an interdisciplinary setting: 1-year prospective cohort. Am J Obstet Gynecol. 2018 Jan;218(1):114.e1-114.e12. doi: 10.1016/j.ajog.2017.10.002. Epub 2017 Oct 12. PMID 29031895
- [Derived] Liu YD, Noga H, Allaire C, Bedaiwy MA, Lee CE, Williams C, Booth A, Galea LAM, Kaida A, Ogilvie GS, Brotto LA, Yong PJ. Mental Health Outcomes of Endometriosis Patients during the COVID-19 Pandemic: Impact of Pre-pandemic Central Nervous System Sensitization. J Pain. 2024 Jul;25(7):104481. doi: 10.1016/j.jpain.2024.01.346. Epub 2024 Jan 19. PMID 38246253
- [Derived] Alfaraj S, Noga H, Allaire C, Williams C, Lisonkova S, Yong PJ, Bedaiwy MA. Negative Sliding Sign during Dynamic Ultrasonography Predicts Low Endometriosis Fertility Index at Laparoscopy. J Minim Invasive Gynecol. 2021 Feb;28(2):249-258.e2. doi: 10.1016/j.jmig.2020.05.003. Epub 2020 May 13. PMID 32416264
- [Derived] Wahl KJ, Orr NL, Lisonek M, Noga H, Bedaiwy MA, Williams C, Allaire C, Albert AY, Smith KB, Cox S, Yong PJ. Deep Dyspareunia, Superficial Dyspareunia, and Infertility Concerns Among Women With Endometriosis: A Cross-Sectional Study. Sex Med. 2020 Jun;8(2):274-281. doi: 10.1016/j.esxm.2020.01.002. Epub 2020 Feb 13. PMID 32061579
- [Derived] Orr NL, Wahl KJ, Noga H, Allaire C, Williams C, Bedaiwy MA, Albert A, Smith KB, Yong PJ. Phenotyping Sexual Pain in Endometriosis Using the Central Sensitization Inventory. J Sex Med. 2020 Apr;17(4):761-770. doi: 10.1016/j.jsxm.2019.12.019. Epub 2020 Jan 24. PMID 31983669
- See also: Endometriosis Pelvic Pain Laboratory — http://yonglab.med.ubc.ca/